CLINICAL TRIAL: NCT06844864
Title: Identification of Adaptive and Trained Immune Mechanisms Driving Tissue Fibrosis in IgG4-Related Disease
Brief Title: Adaptive and Trained Immunity in the Pathogenesis of IgG4-Related Disease
Acronym: TRIM4
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Emanuel Della Torre, Principal Investigator, Assistant Professor of Internal Medicine, IRCCS San Raffaele
Other Study IDs: 2022FH5R92; 2022FH5R92 (Other Grant/Funding Number: Ministero dell'Università e della Ricerca)
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: IgG4 Related Disease
Keywords: Trained immunity
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — peripheral blood to isolate pbmc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Enquire involvement of trained immunity in the pathogenesis of IgG4RD

DETAILED DESCRIPTION:
Enquire involvement of trained immunity in the pathogenesis of IgG4RD using primary macrophages and co-cultures with patient derived fibroblasts. The investigators will first assess whether macrophages from patients are trained compared to macrophages of healthy controls and then challenge them with IgG from IgG4RD patients to evaluate the functional effects on cultivated fibroblasts.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adult subjects > or = 18 years of age
* Subjects capable of providing informed consent
* Active IgG4-RD based on the IgG4-related disease activity index
* Fulfillment of the 2019 ACR/EULAR Classification Criteria for IgG4RD

Healthy Controls:

* Adult subjects > or = 18 years of age
* Subjects capable of providing informed consent

Exclusion Criteria:

Patients and healthy controls:

* Subjects < 18 years of age
* Pregnant women
* Comorbidities (other ongoing active autoimmune diseases, ongoing cancer, ongoing infections)
* Ongoing immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with IgG4-related disease and healthy controls
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of collagen Ia in the supernant of macrophage/fibroblast co-cultures | 7 months
  Concentration of collagen Ia (ng/uL) in the supernant of macrophage/fibroblast co-cultures through ELISA assay

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy